CLINICAL TRIAL: NCT04584736
Title: To Evaluate the Efficacy and Safety of Combination Therapy of Pitavastatin and Ezetimibe Versus Monotherapy of Pitavastatin in Patients With Primary Hypercholesterolemia
Brief Title: To Evaluate the Efficacy and Safety in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JWP-PTZ-301
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2020-08

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — pitavastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Livalo 2mg, Ezetrol 10mg (Experimental): Pitavastatin 2mg, Ezetimibe 10mg
  Interventions: Drug: Livalo, Ezetrol
- Livalo 2mg (Active Comparator): Pitavastatin 2mg
  Interventions: Drug: Livalo, Ezetrol
- Livalo 4mg, Ezetrol 10mg (Experimental): Pitavastatin 4mg, Ezetimibe 10mg
  Interventions: Drug: Livalo, Ezetrol
- Livalo 4mg (Active Comparator): Pitavastatin 4mg
  Interventions: Drug: Livalo, Ezetrol

INTERVENTIONS:
Drug: Livalo, Ezetrol — Pitavastatin+Ezetimibe Pitavastatin
  Other Names: Pitavastatin, Ezetimibe

SUMMARY:
To Evaluate the Efficacy and Safety of Combination Therapy of Pitavastatin and Ezetimibe Versus Monotherapy of Pitavastatin in Patients With Primary Hypercholesterolemia.

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-blinded, Active-controlled, Factorial Design Phase 3 Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hypercholesterolemia

Exclusion Criteria:

* The subject not meet the specified LDL-C level

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
% change in LDL-C level from baseline at Week 8 | Week 8
  change in LDL-C level

SECONDARY OUTCOMES:
Change in LDL-C level from baseline at Week 4 and Week 8 | Week 4 and Week 8
  change in LDL-C level

CONTACTS AND LOCATIONS:
Overall Officials: dongryeong lee, Manager, Study Chair — +82-2-840-6982
Locations (1):
- Gangdong Sacred Heart Hospital, Seoul, Korea, South Korea

REFERENCES:
- [Derived] Jeong HS, Hong SJ, Cho JM, Han KH, Cha DH, Jo SH, Kang HJ, Choi SY, Choi CU, Cho EJ, Jeong YH, Gwon HC, Kim BK, Lee SY, Kim SH, Ahn JC, Hong YJ, Kim WS, Woo SI, Park TH, Han KR. A Multicenter, Randomized, Double-blind, Active-controlled, Factorial Design, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Combination Therapy of Pitavastatin and Ezetimibe Versus Monotherapy of Pitavastatin in Patients With Primary Hypercholesterolemia. Clin Ther. 2022 Oct;44(10):1310-1325. doi: 10.1016/j.clinthera.2022.09.001. Epub 2022 Oct 12. PMID 36241463